CLINICAL TRIAL: NCT01584674
Title: A Prospective Clinical Trial Evaluating the Efficacy of the KLOX Biophotonic System (KLOX KLGA0105-01 and KLOX THERA LAMP) On Moderate to Severe Acne
Brief Title: A Clinical Trial Evaluating the Safety and Efficacy of the KLOX Biophotonic System in Moderate to Severe Acne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KLOX Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-K1005-P001
Record Dates: First submitted 2012-04-19; First posted 2012-04-25 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KLOX Biophotonic System (Experimental): KLOX Biophotonic System (KLOX KLGA0105-01 photo-converter gel and KLOX THERA lamp) will be administered twice a week for 6 weeks followed by a 6-week follow up period
  Interventions: Device: KLOX Biophotonic System
- Control (untreated hemiface) (No Intervention): No treatment will be administered on the control hemiface

INTERVENTIONS:
Device: KLOX Biophotonic System — KLOX Biophotonic System (KLOX KLGA0105-01 photo-converter gel and KLOX THERA lamp) will be administered twice a week for 6 weeks followed by a 6-week follow up period
  Arms: KLOX Biophotonic System

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the KLOX Biophotonic System in patients with moderate to severe facial acne vulgaris using a split-face design (treated hemiface vs untreated hemiface).

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female 16 - 30 years of age.
2. Fitzpatrick skin type I through IV.
3. Known medical history of active acne vulgaris for at least 6 months.
4. Moderate-to-severe facial acne, as defined by:

   Moderate is defined as a patient with an IGA of 3 with 20 to 40 inflammatory lesions (papules and pustules) and no more than 1 nodule. Severe is defined as a patient with an IGA of 4 with a greater than 40 inflammatory lesions with the presence of no more than 2 nodules and/or inflammatory scaring type lesion. Also note that all patients should have a similar disease stage on both sides of their face.
5. The patient must have a clinical examination prior to treatment.
6. The patient must have signed the consent form.
7. The patient must be willing to return for follow-up visits.
8. Females of child bearing potential must have a negative pregnancy test result at baseline and both male and female patients must be willing to adhere to a birth control method.

Exclusion Criteria:

1. Active skin infection on the face. Patient must not have active, localized or systemic infection.
2. Facial aesthetic procedure, including laser therapy and injectables within the last 6 months.
3. Enrollment in another acne study or other dermatological study using light therapy including tanning beds within 120 days of enrollment. Patients must not take part or intend to take part in another study liable to interfere with this study whatever the region of the body considered for 30 days prior to the study start and 30 days following completion of the study.
4. History of head and/or neck irradiation.
5. Use of a hormonal contraception is prohibited unless the birth control has been stable for the past 3 months. Note that patient that are presently taking or have taken in past 30 days Cyproterone Acetate + Ethinyl Estradiol (Diane-35) are not eligible for this study.
6. Any facial dermatological conditions that could hinder or interfere with clinical assessments.
7. Immunosuppression and/or cortisone therapy in the past 4 months.
8. Bleeding diathesis.
9. Medications or supplements affecting coagulation.
10. Isotretinoin within the last 24 weeks.
11. Pregnant, breast-feeding or pregnancy planned during the trial.
12. History of facial nerve palsy or marked facial asymmetry.
13. History of neuromuscular disorder.
14. Prior facial surgery that alters subcutaneous tissues (e.g., rhytidectomy).
15. Use of non-acne topical medication that could interfere with study treatment.
16. Physical or psychiatric condition the investigator deems would preclude participation in the study. (e.g. Polycystic Ovary disease)
17. Unwillingness to refrain from excess sun exposure or tanning beds during the healing process -

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving a total reduction of at least 2 grades in the Investigator's Global Assessment (IGA) scale | 12 weeks

SECONDARY OUTCOMES:
Reduction in inflammatory lesions | 6 and 12 weeks
Proportion of patients achieving a reduction of at least 1 grade in the Investigator's Global Assessment (IGA) scale | 6 and 12 weeks
Proportion of patients achieving a reduction to grade 1 or 0 in the Investigator's Global Assessment (IGA) scale | 6 and 12 weeks
Patient satisfaction questionnaire | 6 and 12 weeks
Pain assessment using a visual analogue scale | 12 weeks
Safety evaluations (treatment-emergent and treatment related adverse events) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Greece (3):
  - Attikon University General Hospital, Athens
  - Andreas Sygros Hospital, Athens
  - Papageorgiou Hospital, Thessaloniki